CLINICAL TRIAL: NCT02261051
Title: Symptom Management, Quality of Life and Satisfaction With Care for Advanced Stage Cancers - Control Arm
Acronym: LCCM-Control
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty in recruitment and change in study site protocols.
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-48
Record Dates: First submitted 2014-09-29; First posted 2014-10-10 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Cancer; Advanced Cancer
Keywords: Palliative Care; Hospice; End of Life; Health Service Utilization; Quality of Life
MeSH Terms: conditions — Neoplasms; Death; Patient Acceptance of Health Care | interventions — Standard of Care

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-concurrent control group: A group of advanced cancer patients who received care at our Center before implementation of the LCCM model. They will receive current standard of care.
  This current study is to collect data on the control group only. After system redesign, we will open an intervention arm study to collect data after implementation of the new care model (about 18-24 months from start of control phase).
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Patients will be cared for using current standard of care preceding the design and implementation of the LCCM model of care.

SUMMARY:
Symptom Management, Quality of Life and Satisfaction with Care for Advanced Stage Cancers is the first part of a two part study (The Lancaster Cancer Care Model (LCCM) - Non-Concurrent Control Study). The primary aim of the study is to compare the proportion of advanced cancer patients who have a hospitalization or emergency department visit in the last 6 months of life before and after implementation of a new care model that provides more comprehensive symptom management and supportive care, including earlier referral to palliative care. The secondary comparative aim is to assess measures of quality of life and satisfaction in both groups. This current study is to collect data on the control group only. After system redesign, we will open an intervention arm study to collect data after implementation of the new care model (about 18-24 months from start of control phase).

DETAILED DESCRIPTION:
Symptom Management, Quality of Life and Satisfaction with Care for Advanced Stage Cancers is the first part of a two part study (The Lancaster Cancer Care Model (LCCM) - Non-Concurrent Control Study) that was submitted to the National Cancer Institute (NCI) for funding. A decision on funding the full study should be forthcoming in the early part of 2015. The primary aim of the study is to compare the proportion of advanced cancer patients who have a hospitalization or emergency department visit in the last 6 months of life before and after implementation of a new care model that provides more comprehensive symptom management and supportive care, including earlier referral to palliative care. The secondary comparative aim is to assess measures of quality of life and satisfaction in both groups. To accomplish the aims of the study by the end of the funding period, we propose to begin data collection in advance of a funding decision. Should the study not receive funding, the data collected will be used to inform decisions regarding other funding applications and/or implementation of program changes at the Ann B. Barshinger Cancer Institute. Data collection does not represent more than minimal risk for the patients enrolled.

This protocol is for the first phase of the study, which is the enrollment and collection of data on the control group, to serve as the baseline for comparison regarding hospitalizations, ED visits, quality of life, and patient and family satisfaction. To achieve sufficient number of subjects and observed deaths in the control group, we are targeting the start of enrollment and data collection in this group during the third quarter of 2014. If the project is funded, the intervention and enrollment in the intervention group are targeted to start in the second quarter of 2016. Background and study aims are presented for the entire project to provide context, but the intent of this application is only for approval of the enrollment and data collection on the control subjects (which contributes to aims 2 and 3 of the larger project). A second protocol would be presented for review and approval at the start of the intervention if the project funding is granted.

In phase one of the project, subjects would be approached and consented at the point of a determination/diagnosis of advanced cancer and followed until the end of life or the start of the intervention period in the 2nd quarter of 2016 (whichever comes first) per protocol.

This current study is to collect data on the control group only. After system redesign, we will open an intervention arm study to collect data after implementation of the new care model (about 18-24 months from start of control phase).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with a solid tumor-type cancer that is considered either advanced and unresectable or metastatic

Exclusion Criteria:

* Non-English speaking
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population includes patients newly diagnosed with a solid tumor-type cancer that is considered either advanced and unresectable or metastatic. Patients also will be at least 18 years of age and English-speaking.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Frequency of patients' ED visits and hospitalizations | Collected at baseline and every 2 months from enrollment until death from any cause or assessed up to 18 months
  All cause: ED admission treat and release, ED admission to inpatient visit and direct inpatient admission

SECONDARY OUTCOMES:
Patient quality of life | Collected at baseline and every 2 months from enrollment until death from any cause or assessed up to 18 months
  Assessed with FACT-G (Functional Assessment of Cancer-General measure)
Patient satisfaction | Collected at baseline and every 2 months from enrollment until death from any cause or assessed up to 18 months
  Assessed with FAMCARE-2 (patient and family satisfaction with care)
Caregiver burden | Collected at baseline and every 2 months from enrollment until death from any cause or assessed up to 18 months
  Assessed with BASC (Brief Assessment Scale for Caregivers) Caregiver Burden
Caregiver satisfaction | Collected at baseline and every 2 months from enrollment until death from any cause or assessed up to 18 months
  Assessed with FAMCARE-2 (patient and family satisfaction with care)
Patient symptoms | Collected at baseline and every outpatient oncology clinic visit from enrollment until death from any cause or assessed up to 18 months
  Assessed with the ESAS-R (Edmonton Symptom Assessment System Revised) and ECOG (Eastern Cooperative Oncology Group) performance status

CONTACTS AND LOCATIONS:
Overall Officials: Shanthi Sivendran, MD, MSCR, Study Director — Lancaster General Ann B. Barshinger Cancer Institute; Randy Oyer, MD, Study Director — Lancaster General Ann B. Barshinger Cancer Institute; Nik Buescher, Principal Investigator — Lancaster General Ann B. Barshinger Cancer Institute; Joan Harrold, MD, Principal Investigator — Palliative Medicine Consultants; Barbara Martin, PhD, Principal Investigator — Lancaster General Research Institute; Kristina Newport, MD, Principal Investigator — Palliative Medicine Consultants; Michael Horst, PhD, Principal Investigator — Lancaster General Research Institute
Locations (1):
- Lancaster General Ann B. Barshinger Cancer Institute, Lancaster, Pennsylvania, United States

REFERENCES:
- [Background] Aoun S, Bird S, Kristjanson LJ, Currow D. Reliability testing of the FAMCARE-2 scale: measuring family carer satisfaction with palliative care. Palliat Med. 2010 Oct;24(7):674-81. doi: 10.1177/0269216310373166. Epub 2010 Jul 9. PMID 20621947
- [Background] Back AL, Arnold RM, Baile WF, Tulsky JA, Fryer-Edwards K. Approaching difficult communication tasks in oncology. CA Cancer J Clin. 2005 May-Jun;55(3):164-77. doi: 10.3322/canjclin.55.3.164. PMID 15890639
- [Background] Baile WF, Lenzi R, Parker PA, Buckman R, Cohen L. Oncologists' attitudes toward and practices in giving bad news: an exploratory study. J Clin Oncol. 2002 Apr 15;20(8):2189-96. doi: 10.1200/JCO.2002.08.004. PMID 11956281
- [Background] Bakitas M, Lyons KD, Hegel MT, Balan S, Brokaw FC, Seville J, Hull JG, Li Z, Tosteson TD, Byock IR, Ahles TA. Effects of a palliative care intervention on clinical outcomes in patients with advanced cancer: the Project ENABLE II randomized controlled trial. JAMA. 2009 Aug 19;302(7):741-9. doi: 10.1001/jama.2009.1198. PMID 19690306
- [Background] Barnato AE, Llewellyn-Thomas HA, Peters EM, Siminoff L, Collins ED, Barry MJ. Communication and decision making in cancer care: setting research priorities for decision support/patients' decision aids. Med Decis Making. 2007 Sep-Oct;27(5):626-34. doi: 10.1177/0272989X07306788. Epub 2007 Sep 14. PMID 17873249
- [Background] Brumley RD, Enguidanos S, Cherin DA. Effectiveness of a home-based palliative care program for end-of-life. J Palliat Med. 2003 Oct;6(5):715-24. doi: 10.1089/109662103322515220. PMID 14622451
- [Background] Brumley R, Enguidanos S, Jamison P, Seitz R, Morgenstern N, Saito S, McIlwane J, Hillary K, Gonzalez J. Increased satisfaction with care and lower costs: results of a randomized trial of in-home palliative care. J Am Geriatr Soc. 2007 Jul;55(7):993-1000. doi: 10.1111/j.1532-5415.2007.01234.x. PMID 17608870
- [Background] Bull JH, Whitten E, Morris J, Hooper RN, Wheeler JL, Kamal A, Abernethy AP. Demonstration of a sustainable community-based model of care across the palliative care continuum. J Pain Symptom Manage. 2012 Dec;44(6):797-809. doi: 10.1016/j.jpainsymman.2011.12.278. Epub 2012 Jul 7. PMID 22771124
- [Background] Carter GL, Lewin TJ, Gianacas L, Clover K, Adams C. Caregiver satisfaction with out-patient oncology services: utility of the FAMCARE instrument and development of the FAMCARE-6. Support Care Cancer. 2011 Apr;19(4):565-72. doi: 10.1007/s00520-010-0858-1. Epub 2010 Mar 28. PMID 20349317
- [Background] Cheifetz O, Packham TL, Macdermid JC. Rasch analysis of the Edmonton Symptom Assessment System and research implications. Curr Oncol. 2014 Apr;21(2):e186-94. doi: 10.3747/co.21.1735. PMID 24764703
- [Background] Colon M. Hospice and Latinos: a review of the literature. J Soc Work End Life Palliat Care. 2005;1(2):27-43. doi: 10.1300/J457v01n02_04. PMID 17387062
- [Background] Conrad KJ, Iris M, Ridings JW, Langley K, Wilber KH. Self-report measure of financial exploitation of older adults. Gerontologist. 2010 Dec;50(6):758-73. doi: 10.1093/geront/gnq054. Epub 2010 Jul 28. PMID 20667945
- [Background] Daugherty CK, Hlubocky FJ. What are terminally ill cancer patients told about their expected deaths? A study of cancer physicians' self-reports of prognosis disclosure. J Clin Oncol. 2008 Dec 20;26(36):5988-93. doi: 10.1200/JCO.2008.17.2221. Epub 2008 Nov 24. PMID 19029419
- [Background] de Kock I, Mirhosseini M, Lau F, Thai V, Downing M, Quan H, Lesperance M, Yang J. Conversion of Karnofsky Performance Status (KPS) and Eastern Cooperative Oncology Group Performance Status (ECOG) to Palliative Performance Scale (PPS), and the interchangeability of PPS and KPS in prognostic tools. J Palliat Care. 2013 Autumn;29(3):163-9. PMID 24380215
- [Background] Degenholtz HB, Thomas SB, Miller MJ. Race and the intensive care unit: disparities and preferences for end-of-life care. Crit Care Med. 2003 May;31(5 Suppl):S373-8. doi: 10.1097/01.CCM.0000065121.62144.0D. No abstract available. PMID 12771586
- [Background] Doll KM, Stine JE, Van Le L, Moore DT, Bae-Jump V, Brewster WR, Soper JT, Boggess JF, Gehrig PA, Kim KH. Outpatient end of life discussions shorten hospital admissions in gynecologic oncology patients. Gynecol Oncol. 2013 Jul;130(1):152-5. doi: 10.1016/j.ygyno.2013.03.020. Epub 2013 Mar 29. PMID 23542684
- [Background] El-Jawahri A, Greer JA, Temel JS. Does palliative care improve outcomes for patients with incurable illness? A review of the evidence. J Support Oncol. 2011 May-Jun;9(3):87-94. doi: 10.1016/j.suponc.2011.03.003. PMID 21702398
- [Background] Enguidanos S, Housen P, Goldstein R, Vesper E, Allen J, Braun W. Physician and nurse perceptions of a new inpatient palliative care consultation project: implications for education and training. J Palliat Med. 2009 Dec;12(12):1137-42. doi: 10.1089/jpm.2009.0131. PMID 19708839
- [Background] Gade G, Venohr I, Conner D, McGrady K, Beane J, Richardson RH, Williams MP, Liberson M, Blum M, Della Penna R. Impact of an inpatient palliative care team: a randomized control trial. J Palliat Med. 2008 Mar;11(2):180-90. doi: 10.1089/jpm.2007.0055. PMID 18333732
- [Background] Glajchen M, Kornblith A, Homel P, Fraidin L, Mauskop A, Portenoy RK. Development of a brief assessment scale for caregivers of the medically ill. J Pain Symptom Manage. 2005 Mar;29(3):245-54. doi: 10.1016/j.jpainsymman.2004.06.017. PMID 15781175
- [Background] Glare PA, Semple D, Stabler SM, Saltz LB. Palliative care in the outpatient oncology setting: evaluation of a practical set of referral criteria. J Oncol Pract. 2011 Nov;7(6):366-70. doi: 10.1200/JOP.2011.000367. PMID 22379418
- [Background] Greer JA, Pirl WF, Jackson VA, Muzikansky A, Lennes IT, Heist RS, Gallagher ER, Temel JS. Effect of early palliative care on chemotherapy use and end-of-life care in patients with metastatic non-small-cell lung cancer. J Clin Oncol. 2012 Feb 1;30(4):394-400. doi: 10.1200/JCO.2011.35.7996. Epub 2011 Dec 27. PMID 22203758
- [Background] Hui D, Elsayem A, De la Cruz M, Berger A, Zhukovsky DS, Palla S, Evans A, Fadul N, Palmer JL, Bruera E. Availability and integration of palliative care at US cancer centers. JAMA. 2010 Mar 17;303(11):1054-61. doi: 10.1001/jama.2010.258. PMID 20233823
- [Background] The future of nursing: the Institute of Medicine (IOM) issues report. The future of nursing: leading change, advancing health. Prairie Rose. 2010 Nov-2011 Jan;79(4):6. No abstract available. PMID 21207799
- [Background] Jacobsen J, Jackson V, Dahlin C, Greer J, Perez-Cruz P, Billings JA, Pirl W, Temel J. Components of early outpatient palliative care consultation in patients with metastatic nonsmall cell lung cancer. J Palliat Med. 2011 Apr;14(4):459-64. doi: 10.1089/jpm.2010.0382. Epub 2011 Mar 18. PMID 21417739
- [Background] Keating NL, Landrum MB, Rogers SO Jr, Baum SK, Virnig BA, Huskamp HA, Earle CC, Kahn KL. Physician factors associated with discussions about end-of-life care. Cancer. 2010 Feb 15;116(4):998-1006. doi: 10.1002/cncr.24761. PMID 20066693
- [Background] Little RJ, D'Agostino R, Cohen ML, Dickersin K, Emerson SS, Farrar JT, Frangakis C, Hogan JW, Molenberghs G, Murphy SA, Neaton JD, Rotnitzky A, Scharfstein D, Shih WJ, Siegel JP, Stern H. The prevention and treatment of missing data in clinical trials. N Engl J Med. 2012 Oct 4;367(14):1355-60. doi: 10.1056/NEJMsr1203730. No abstract available. PMID 23034025
- [Background] Meier DE, Beresford L. Outpatient clinics are a new frontier for palliative care. J Palliat Med. 2008 Jul;11(6):823-8. doi: 10.1089/jpm.2008.9886. No abstract available. PMID 18715171
- [Background] Milne D, Aranda S, Jefford M, Schofield P. Development and validation of a measurement tool to assess perceptions of palliative care. Psychooncology. 2013 Apr;22(4):940-6. doi: 10.1002/pon.3071. Epub 2012 Mar 27. PMID 22451082
- [Background] Morden NE, Chang CH, Jacobson JO, Berke EM, Bynum JP, Murray KM, Goodman DC. End-of-life care for Medicare beneficiaries with cancer is highly intensive overall and varies widely. Health Aff (Millwood). 2012 Apr;31(4):786-96. doi: 10.1377/hlthaff.2011.0650. PMID 22492896
- [Background] Morrison RS, Augustin R, Souvanna P, Meier DE. America's care of serious illness: a state-by-state report card on access to palliative care in our nation's hospitals. J Palliat Med. 2011 Oct;14(10):1094-6. doi: 10.1089/jpm.2011.9634. Epub 2011 Sep 16. No abstract available. PMID 21923412
- [Background] Morrison RS, Dietrich J, Ladwig S, Quill T, Sacco J, Tangeman J, Meier DE. Palliative care consultation teams cut hospital costs for Medicaid beneficiaries. Health Aff (Millwood). 2011 Mar;30(3):454-63. doi: 10.1377/hlthaff.2010.0929. PMID 21383364
- [Background] Muir JC, Daly F, Davis MS, Weinberg R, Heintz JS, Paivanas TA, Beveridge R. Integrating palliative care into the outpatient, private practice oncology setting. J Pain Symptom Manage. 2010 Jul;40(1):126-35. doi: 10.1016/j.jpainsymman.2009.12.017. PMID 20619215
- [Background] O'Mahony S, McHenry J, Snow D, Cassin C, Schumacher D, Selwyn PA. A review of barriers to utilization of the medicare hospice benefits in urban populations and strategies for enhanced access. J Urban Health. 2008 Mar;85(2):281-90. doi: 10.1007/s11524-008-9258-y. PMID 18240022
- [Background] Oechsle K, Goerth K, Bokemeyer C, Mehnert A. Anxiety and depression in caregivers of terminally ill cancer patients: impact on their perspective of the patients' symptom burden. J Palliat Med. 2013 Sep;16(9):1095-101. doi: 10.1089/jpm.2013.0038. Epub 2013 Aug 3. PMID 23909373
- [Background] Pantilat SZ, Kerr KM, Billings JA, Bruno KA, O'Riordan DL. Palliative care services in California hospitals: program prevalence and hospital characteristics. J Pain Symptom Manage. 2012 Jan;43(1):39-46. doi: 10.1016/j.jpainsymman.2011.03.021. Epub 2011 Jul 30. PMID 21802898
- [Background] Park CM, Koh Y, Jeon K, Na S, Lim CM, Choi WI, Lee YJ, Kim SC, Chon GR, Kim JH, Kim JY, Lim J, Rhee CK, Park S, Kim HC, Lee JH, Lee JH, Park J, Cho J, Koh SO, Suh GY; Validation of Simplified acute physiology score 3 in Korean Intensive care unit (VSKI) study group; Korean Study Group on Respiratory Failure (KOSREF). Impact of Eastern Cooperative Oncology Group Performance Status on hospital mortality in critically ill patients. J Crit Care. 2014 Jun;29(3):409-13. doi: 10.1016/j.jcrc.2014.01.016. Epub 2014 Jan 30. PMID 24603001
- [Background] Peppercorn JM, Smith TJ, Helft PR, Debono DJ, Berry SR, Wollins DS, Hayes DM, Von Roenn JH, Schnipper LE; American Society of Clinical Oncology. American society of clinical oncology statement: toward individualized care for patients with advanced cancer. J Clin Oncol. 2011 Feb 20;29(6):755-60. doi: 10.1200/JCO.2010.33.1744. Epub 2011 Jan 24. PMID 21263086
- [Background] Pereira J, Green E, Molloy S, Dudgeon D, Howell D, Krzyzanowska MK, Mahase W, Tabing R, Urowitz S, Macdougall L. Population-based standardized symptom screening: Cancer Care Ontario's Edmonton Symptom Assessment System and performance status initiatives. J Oncol Pract. 2014 May;10(3):212-4. doi: 10.1200/JOP.2014.001390. Epub 2014 Apr 22. No abstract available. PMID 24756143
- [Background] Prince-Paul M, Burant CJ, Saltzman JN, Teston LJ, Matthews CR. The effects of integrating an advanced practice palliative care nurse in a community oncology center: a pilot study. J Support Oncol. 2010 Jan-Feb;8(1):21-7. PMID 20235420
- [Background] Quill TE, Abernethy AP. Generalist plus specialist palliative care--creating a more sustainable model. N Engl J Med. 2013 Mar 28;368(13):1173-5. doi: 10.1056/NEJMp1215620. Epub 2013 Mar 6. No abstract available. PMID 23465068
- [Background] Rabow MW, Dibble SL, Pantilat SZ, McPhee SJ. The comprehensive care team: a controlled trial of outpatient palliative medicine consultation. Arch Intern Med. 2004 Jan 12;164(1):83-91. doi: 10.1001/archinte.164.1.83. PMID 14718327
- [Background] Ramey SJ, Chin SH. Disparity in hospice utilization by African American patients with cancer. Am J Hosp Palliat Care. 2012 Aug;29(5):346-54. doi: 10.1177/1049909111423804. Epub 2011 Oct 23. PMID 22025746
- [Background] Rogers M, Todd C. Information exchange in oncology outpatient clinics: source, valence and uncertainty. Psychooncology. 2002 Jul-Aug;11(4):336-45. doi: 10.1002/pon.575. PMID 12203746
- [Background] Scheffey C, Kestenbaum MG, Wachterman MW, Connor SR, Fine PG, Davis MS, Muir JC. Clinic-based outpatient palliative care before hospice is associated with longer hospice length of service. J Pain Symptom Manage. 2014 Oct;48(4):532-9. doi: 10.1016/j.jpainsymman.2013.10.017. Epub 2014 Mar 27. PMID 24680626
- [Background] Schenker Y, Crowley-Matoka M, Dohan D, Rabow MW, Smith CB, White DB, Chu E, Tiver GA, Einhorn S, Arnold RM. Oncologist factors that influence referrals to subspecialty palliative care clinics. J Oncol Pract. 2014 Mar;10(2):e37-44. doi: 10.1200/JOP.2013.001130. Epub 2013 Dec 3. PMID 24301842
- [Background] Smith TJ, Hillner BE. Bending the cost curve in cancer care. N Engl J Med. 2011 May 26;364(21):2060-5. doi: 10.1056/NEJMsb1013826. No abstract available. PMID 21612477
- [Background] Smith TJ, Temin S, Alesi ER, Abernethy AP, Balboni TA, Basch EM, Ferrell BR, Loscalzo M, Meier DE, Paice JA, Peppercorn JM, Somerfield M, Stovall E, Von Roenn JH. American Society of Clinical Oncology provisional clinical opinion: the integration of palliative care into standard oncology care. J Clin Oncol. 2012 Mar 10;30(8):880-7. doi: 10.1200/JCO.2011.38.5161. Epub 2012 Feb 6. PMID 22312101
- [Background] Sprandio JD. Oncology patient-centered medical home. J Oncol Pract. 2012 May;8(3 Suppl):47s-9s. doi: 10.1200/JOP.2012.000590. PMID 22942826
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076
- [Background] Storey CP Jr. Why oncologists should refer patients earlier for hospice care. Oncology (Williston Park). 2011 Nov 30;25(13):1285. No abstract available. PMID 22272500
- [Background] Stubenrauch JM. Rectal cancer rates rising in patients under 40. Am J Nurs. 2010 Nov;110(11):15. doi: 10.1097/01.NAJ.0000390504.69533.e3. No abstract available. PMID 20980880
- [Background] Tavernier SS. Translating research on the distress thermometer into practice. Clin J Oncol Nurs. 2014;18 Suppl:26-30. doi: 10.1188/14.CJON.S1.26-30. PMID 24480660
- [Background] Temel JS, Greer JA, Admane S, Gallagher ER, Jackson VA, Lynch TJ, Lennes IT, Dahlin CM, Pirl WF. Longitudinal perceptions of prognosis and goals of therapy in patients with metastatic non-small-cell lung cancer: results of a randomized study of early palliative care. J Clin Oncol. 2011 Jun 10;29(17):2319-26. doi: 10.1200/JCO.2010.32.4459. Epub 2011 May 9. PMID 21555700
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Von Roenn JH, Temel J. The integration of palliative care and oncology: the evidence. Oncology (Williston Park). 2011 Nov 30;25(13):1258-60, 1262, 1264-5. PMID 22272492
- [Background] Walshe C, Todd C, Caress A, Chew-Graham C. Patterns of access to community palliative care services: a literature review. J Pain Symptom Manage. 2009 May;37(5):884-912. doi: 10.1016/j.jpainsymman.2008.05.004. Epub 2008 Dec 21. PMID 19097748
- [Background] Wright AA, Zhang B, Ray A, Mack JW, Trice E, Balboni T, Mitchell SL, Jackson VA, Block SD, Maciejewski PK, Prigerson HG. Associations between end-of-life discussions, patient mental health, medical care near death, and caregiver bereavement adjustment. JAMA. 2008 Oct 8;300(14):1665-73. doi: 10.1001/jama.300.14.1665. PMID 18840840
- [Background] Zhang B, Wright AA, Huskamp HA, Nilsson ME, Maciejewski ML, Earle CC, Block SD, Maciejewski PK, Prigerson HG. Health care costs in the last week of life: associations with end-of-life conversations. Arch Intern Med. 2009 Mar 9;169(5):480-8. doi: 10.1001/archinternmed.2008.587. PMID 19273778
- See also: Cancer Facts and Figures 2014. (n.d.). Retrieved May 21, 2014, from http://www.cancer.org/acs/groups/content/@research/documents/webcontent/acspc-042151.pdf — http://www.cancer.org/acs/groups/content/@research/documents/webcontent/acspc-042151.pdf
- See also: National Community Cancer Centers Program Pilot Fact Sheet, 2007-2010. (n.d.) Retrieved June 16, 2014 from http://ncccp.cancer.gov/Media/FactSheet.htm — http://ncccp.cancer.gov/Media/FactSheet.htm